CLINICAL TRIAL: NCT04245618
Title: Role of Neoadjuvant Chemotherapy in the Conservative Management of Non-muscle Invasive Bladder Cancer (NMIBC) T1b
Brief Title: Neoadjuvant Chemotherapy in Non Muscle Invasive T1b Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, heba mahmoud mohamed, principal investigator, Assiut University
Other Study IDs: NAC in T1 Bladder cancer
Record Dates: First submitted 2020-01-26; First posted 2020-01-29 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: neoadjuvant chemotherapy ( cisplatin - gemcitabine) — Neoadjuvant chemotherapy before TURBT
  Other Names: cisplatin - gemzar

SUMMARY:
The aim of our study is to evaluate the benefit of NAC in T1b NMIBC .

DETAILED DESCRIPTION:
Bladder cancer (BC) is the most common malignancy of the urinary tract and the fourth most frequent cancer in the United States, with 79,030 new cases and 16,870 deaths estimated for 2017.

The most common presenting symptom is hematuria, which occurs in about 85% of patients. Hematuria is typically intermittent, gross, and painless. Bladder irritability, usually presenting as urinary frequency, urgency, and dysuria, occurs in about 20% of patients.

Initial diagnostic workup usually involves cystoscopy and urine cytology. Cystoscopy is the gold standard for the initial diagnosis and staging of bladder cancer. If a bladder mass is detected, a transurethral resection of the bladder tumor (TURBT) is performed for full primary tumor staging. The resected bladder tumor specimen should include muscle to fully assess the depth of tumor invasion. If carcinoma in situ (CIS) is detected, multiple random biopsies, including several different areas of the bladder and the prostatic urethra, may be required to assess the extent of involvement.

Abdominal imaging with either CT or MRI is recommended in patients with a high-grade tumor or muscle invasive disease to assess for local lymph node involvement, loco regional extent of disease and the presence of hydronephrosis.

Approximately 75% of patients with urothelial carcinoma of the bladder present with non-muscle-invasive bladder cancer (NMIBC), either confined to the mucosa (Ta and carcinoma in situ [CIS]) or invading the lamina propria (T1) . Clinical T1 high-grade (cT1HG) NMIBC has the highest rate of local recurrence and carries a significant risk of disease progression, clinical understaging, and death from urothelial carcinoma (UC) . The standard of care for adequately resected cT1HG NMIBC is intravesical Bacillus Calmette-Guerin (BCG) with early radical cystectomy (RC) for recurrent or refractory cT1HG disease Pathological upstaging to pathological tumor -2( pT2) is reported in approximately 50% when muscularis propria is absent from the original biopsy, and up to 25% will have lymph node (LN) metastases , which significantly increases the risk for cancer-specific death . These observations imply that a subset of patients with NMIBC that invades into the lamina propria is at a higher risk for clinical understaging and death from UC and may benefit from more aggressive therapy.

Long-term surveillance thus remains the cornerstone of long-term management, and cystoscopy has represented the gold standard modality for over 80 years.

Cisplatin- Gemcitabine (CG) neoadjuvant chemotherapy (NAC) provides pathological downstaging and improved overall survival (OS) for patients with muscle-invasive bladder cancer (MIBC) undergoing RC.

Chemotherapy administered in a neoadjuvant setting comes with some advantages: the ability to deliver effective systemic therapy while the burden of micrometastatic disease is low and is given in a setting in which the patient's performance status is optimal (patient more fit, no loss of renal function, eligibility to optimal cisplatin-based chemotherapy regimens).

High risk features (HRFs) in NMIBC were defined as follows: lymph-vascular invasion (LVI), thickening or induration on Examination under anesthesia( EUA) , tumor-associated hydronephrosis, and variant histology. Tumors with a primary urothelial component and presence of micropapillary, squamous, sarcomatoid, nested variant, glandular, plasmacytoid, adenocarcinoma, or lymphoepithelioma components were classified as tumors of variant histology ( ,also T1b substage has bad prognosis.

The investigators hypothesized that similar high-risk features (HRFs) might identify a high-risk subset of UC patients that could benefit from NAC in the absence of evidence for muscle invasion.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who are older than 18 years old.
2. Histologically confirmed to have Non-muscle invasive bladder cancer, T1bN0M0 ,clinically and radiologically confirmed to have bladder cancer.
3. Patient should have Eastern Cooperative Oncology Group performances status (ECOG)0-1 with adequate hematologic, hepatic and renal functions including hemoglobin>10 /dl, absolute neutrophil count ≥1,500/mm3, platelets ≥100,000/mm3, serum bilirubin <2 mg/dl ,both Alanine transaminase( ALT) and aspartate aminotransferase( AST) ≤2× upper limit of normal (ULN), alkaline phosphates ≤5×ULN,and serum creatinine ≤1.5 mg/dl or creatinine clearance ≥60 ml/min.

Exclusion Criteria:

1. Patients with radiographic evidence of nodal or distant metastases.
2. A past history of upper tract disease, neuroendocrine features.
3. Non-cisplatin-based NAC .
4. Prior radiation therapy to their pelvis.
5. A palpable three-dimensional mass on EUA.
6. Known to be stage 0, T1a, II, III, IV.
7. Active serious infection, or a psychiatric illness that would preclude obtaining informed consent or history of cardiac disease will be excluded.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years confirmed to have T1b Non muscle invasive bladder cancer by biopsy will take neoadjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the benefit of NAC in T1b NMIBC . | baseline
  assessment of the response in correlation with high risk features.

SECONDARY OUTCOMES:
Overall survival (OS) and disease-specific survival (DSS). | 2 years
  Overall survival (OS) and disease-specific survival (DSS).

CONTACTS AND LOCATIONS:
Overall Officials: hoda essa, professor, Study Director — Assiut University

REFERENCES:
- [Background] Cambier S, Sylvester RJ, Collette L, Gontero P, Brausi MA, van Andel G, Kirkels WJ, Silva FC, Oosterlinck W, Prescott S, Kirkali Z, Powell PH, de Reijke TM, Turkeri L, Collette S, Oddens J. EORTC Nomograms and Risk Groups for Predicting Recurrence, Progression, and Disease-specific and Overall Survival in Non-Muscle-invasive Stage Ta-T1 Urothelial Bladder Cancer Patients Treated with 1-3 Years of Maintenance Bacillus Calmette-Guerin. Eur Urol. 2016 Jan;69(1):60-9. doi: 10.1016/j.eururo.2015.06.045. Epub 2015 Jul 23. PMID 26210894
- [Background] Tarin TV, Power NE, Ehdaie B, Sfakianos JP, Silberstein JL, Savage CJ, Sjoberg D, Dalbagni G, Bochner BH. Lymph node-positive bladder cancer treated with radical cystectomy and lymphadenectomy: effect of the level of node positivity. Eur Urol. 2012 May;61(5):1025-30. doi: 10.1016/j.eururo.2012.01.049. Epub 2012 Feb 7. PMID 22342773
- [Background] Chahal R, Harrison SC. Re: an interval longer than 12 weeks between the diagnosis of muscle invasion and cystectomy is associated with worse outcome in bladder carcinoma. J Urol. 2003 Oct;170(4 Pt 1):1327; author reply 1327. No abstract available. PMID 14515867
- [Background] Black PC, Brown GA, Dinney CP. The impact of variant histology on the outcome of bladder cancer treated with curative intent. Urol Oncol. 2009 Jan-Feb;27(1):3-7. doi: 10.1016/j.urolonc.2007.07.010. Epub 2008 Jan 14. PMID 18367107
- [Background] Otto W, van Rhijn BW, Breyer J, Bertz S, Eckstein M, Mayr R, Lausenmeyer EM, Denzinger S, Burger M, Hartmann A. Infiltrative lamina propria invasion pattern as an independent predictor for cancer-specific and overall survival of instillation treatment-naive stage T1 high-grade urothelial bladder cancer. Int J Urol. 2018 May;25(5):442-449. doi: 10.1111/iju.13532. Epub 2018 Feb 22. PMID 29473226
- [Background] Babjuk M, Burger M, Comperat EM, Gontero P, Mostafid AH, Palou J, van Rhijn BWG, Roupret M, Shariat SF, Sylvester R, Zigeuner R, Capoun O, Cohen D, Escrig JLD, Hernandez V, Peyronnet B, Seisen T, Soukup V. European Association of Urology Guidelines on Non-muscle-invasive Bladder Cancer (TaT1 and Carcinoma In Situ) - 2019 Update. Eur Urol. 2019 Nov;76(5):639-657. doi: 10.1016/j.eururo.2019.08.016. Epub 2019 Aug 20. PMID 31443960
- [Background] Martin-Doyle W, Leow JJ, Orsola A, Chang SL, Bellmunt J. Improving selection criteria for early cystectomy in high-grade t1 bladder cancer: a meta-analysis of 15,215 patients. J Clin Oncol. 2015 Feb 20;33(6):643-50. doi: 10.1200/JCO.2014.57.6967. Epub 2015 Jan 5. PMID 25559810
- [Background] Yoshida S, Koga F, Kobayashi S, Ishii C, Tanaka H, Tanaka H, Komai Y, Saito K, Masuda H, Fujii Y, Kawakami S, Kihara K. Role of diffusion-weighted magnetic resonance imaging in predicting sensitivity to chemoradiotherapy in muscle-invasive bladder cancer. Int J Radiat Oncol Biol Phys. 2012 May 1;83(1):e21-7. doi: 10.1016/j.ijrobp.2011.11.065. Epub 2012 Mar 11. PMID 22414281